CLINICAL TRIAL: NCT05593705
Title: The Prevalence of Variations in Attachment and Morphology of Maxillary Labial Frenum on A Sample of Adult Egyptian Population
Brief Title: The Prevalence of Variations in Attachment and Morphology of Labial MLF on A Sample of Adult Egyptian Population
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abeer Ali Hussein Al-Fkih, principal investigator, Cairo University
Other Study IDs: variations in MLF
Record Dates: First submitted 2022-10-09; First posted 2022-10-25 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Labial Tie
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observation — photograph for maxillary labial frenum and measurements with a periodontal probe

SUMMARY:
The study aims at determining the prevalence of the various types of Maxillary Labial Frenum attachment and morphology among adult Egyptian dental outpatients attending the diagnostic center at Faculty of Dentistry, Cairo University.

DETAILED DESCRIPTION:
A frenum is a fibrous band of tissue attached to the bone of the maxilla and mandible, it is frequently superficial to the muscle attachments. There are different types of frena in a normal oral cavity, most notably the maxillary labial frenum, the mandibular labial frenum, the buccal frenum and the lingual frenum. The primary function of frenum is to provide stability of the upper and lower lip. Labial frenal attachments are thin folds of mucous membrane with enclosed muscle fibers originating from orbicularis oris muscle of the upper lip that attaches at the lips to the alveolar mucosa and underlying periosteum on the middle part of the upper lip between the upper central incisors. The labial frenum has unpredictable variation in reference to size, shape, and position during different time periods of growth and development. During the growth period, it is of less clinical importance as it has the ability to decrease in size. At a younger age frenum is generally wide and thick, with time it becomes thin and small .

Abnormal frenum attachment can lead to distension of the gingival sulcus because of frenal pull causing severe periodontal pockets as there is increase plaque accumulation and gingival recession may be caused by the frenum when attached too closely to the gingival margin. It may even affect denture fit or retention. Abnormal labial frenum has also been associated with various syndromes like Ehlers-Danlos syndrome. There are different types and variations of the labial frenum, for this the frenum assessment during oral examination is important in order to avoid misdiagnosis of normal variations as abnormal frenum.

ELIGIBILITY:
Inclusion Criteria:

1. Adult Egyptian patients whose age is above 18 years old.
2. Patient consulting in the outpatient clinic
3. Provide informed consent.

Exclusion Criteria:

1. Patients who have had any orofacial anomalies.
2. Trauma/injuries in the premaxillary region.
3. History of prior orthognathic/frenal surgeries.
4. Missing of one or both central incisors.
5. Patient under any medication known to affect the gingiva (e.g., phenytoin).
6. Syndromes associated with different frenal attachments:

   * Ehlers Danlos syndrome.
   * Infantile hypertrophic pyloric stenosis.
   * Holoprosencephaly.
   * Ellis van Creveld syndrome.
   * Oro facial digital syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Dental patients will be recruited in a consecutive manner from the outpatient Diagnostic center, Faculty of Dentistry, Cairo University.
Sampling Method: Non-Probability Sample
Enrollment: 384 (Estimated)
Dates: Start 2022-11-10 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Prevalence of variations of maxillary labial frenum attachment | through study completion, an average of 1 year
  The primary outcome of the study is the prevalence of variations of maxillary labial frenum attachment. It will be diagnosed by proper history and clinical examination.
  The clinical examination will be performed, patients will be examine lying in a supine position using direct visual method on the dental unit. Under adequate light the upper lip will gently lift with the index finger and thumb of both hands. The site of attachment of frenum will be examined through direct visual examination and intraoral photographs will be also taken. The clinical classification of maxillary frenum insertion by (Mirko, Miroslav and Lubor, 1974)

SECONDARY OUTCOMES:
Morphological labial frenum variations | through study completion, an average of 1 year
  Under adequate light the upper lip will gently lift with the index finger and thumb of both hands. The morphology of frenum will be examined through direct visual examination and intraoral photographs will be also taken. The classification of the frenum variations in morphology are eight different types, simple, persistent tectolabial, simple with appendix, simple with nodule, double frenum, frenum with nichum, bifid frenum and frenum with one or more variation of the above (Sewerin, 1971)

OTHER OUTCOMES:
Papilla presence | through study completion, an average of 1 year
  Assessing the positional relationship among the papilla, cementoenamel junction (CEJ) and adjacent teeth (Cardaropoli, Re and Corrente, 2004)
Gingival Recession Depth (RD) | through study completion, an average of 1 year
  The evaluation will be performed on both frontal and lateral sites using University of North Carolina-15 (UNC 15) probe, and a dental explorer, two variables will be considered: CEJ and cervical discrepancies. Assessment of gingival recession at both buccal and interproximal sites (Cairo et al., 2011)
Midline diastema | through study completion, an average of 1 year
  Visual examination to assess the presence or absence of midline diastema, the "blanch test" use to evaluate the continuity of the tissue fibres of the labial frenum through the diastema to the palatine papilla. The test is accomplished by lifting the upper lip upward and forward until the frenum is tightly stretched. If the procedure produces a blanching or change of contour in this area, the frenum is considered abnormal (Angle, 1907)
Width of keratinized gingiva | through study completion, an average of 1 year
  Measure at the midbuccal aspect of the tooth by University of North Carolina-15 (UNC-15) probe which is color-coded at every millimetre demarcation. The measurement will be from the gingival margin to the mucogingival junction. The mucogingival junction will be identified by the rolling technique, where in the mucosa rolled until the non-movable portion of the attached keratinized tissue is seen (Mazzocco et al., 2011)
Plaque index | through study completion, an average of 1 year
  Teeth in each quadrant will be dried with a blast of air, and presence of visible dental plaque and supragingival calculus will be recorded. Scores 0,1,2,3 (Silness and Löe, 1964), each of the four surfaces of the teeth (buccal, lingual, mesial and distal) is given a score from 0-3. The scores from the four areas of the tooth are added and divided by four in order to give the plaque index for the tooth with the following scores and criteria
Bleeding on Probing | through study completion, an average of 1 year
  Gingival bleeding will be assessed. Gentle probing of the orifice of the gingival crevice. The periodontal probe will be inserted into the gingival sulcus starting at one interproximal area and moving to the other. If bleeding occurs within 10 seconds a positive finding is recorded (Ainamo and Bay, 1975)

IPD SHARING:
Plan to Share IPD: No